CLINICAL TRIAL: NCT02955433
Title: The Impact of Rideshare Transportation Services on Appointment Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Lyft, Inc. (Unknown)
Responsible Party: Principal Investigator, David Grande, Assistant Professor of Medicine at the Perelman School of Medicine, University of Pennsylvania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-824715
Record Dates: First submitted 2016-10-31; First posted 2016-11-04 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Appointments and Schedules; Social Determinants of Health; Transportation; Primary Health Care
Keywords: Rideshare; Digital transportation network; Missed appointment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rideshare (Experimental): The intervention arm will receive an appointment reminder and free transportation for one appointment to travel between the patient's home and primary care clinic using a rideshare-based transportation service.
  Interventions: Other: Rideshare-based transportation
- Control (No Intervention): The control arm will receive an appointment reminder, but no free transportation offer.

INTERVENTIONS:
Other: Rideshare-based transportation
  Other Names: Digital transportation network; Lyft
  Arms: Rideshare

SUMMARY:
This study is a prospective clinical trial designed to primarily test the impact of rideshare-based transportation services from a digital transportation network, Lyft, on reducing primary care clinic missed appointments--a composite outcome of no-shows and same day cancellations--for Medicaid patients. The study population consists of West Philadelphia residents who are established patients at two of the Penn Medicine Primary Care Practices within the University of Pennsylvania Health System. The study subjects are allocated into the intervention or control arm using a pseudorandomization approach - those receiving an appointment reminder on an even calendar day are in the intervention arm and odd calendar day calls are in the control arm.

Secondary outcomes include the time of arrival to the clinics relative to actual appointment time (both arms), prospective utilization of acute care settings (both arms), prospective utilization of primary care (both arms), and description of programmatic metrics in the intervention arm (travel time, misuse, and costs). The investigators will assess the patient experience after each ride using a telephone-based survey and in-depth interviews. All adults with established primary care at the Penn Medicine Clinics, who have Medicaid, and do not require wheelchair accessible rides will be eligible for the rideshare service. The investigators hypothesize that individuals offered a rideshare-based transportation service will have a decreased proportion of missed appointments and same day cancellations as those not offered the service.

ELIGIBILITY:
Inclusion Criteria:

* Patients insured by Medicaid
* Established primary care patient at the Penn Medicine Clinics
* Address in West Philadelphia zip code

Exclusion Criteria:

* Requiring wheelchair accessible transportation. We are unable to guarantee vehicles that will be able to accommodate these patients' physical needs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 786 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
The proportion of missed appointments (no-shows and same-day cancellation) in the intervention arm and the control arm | Within 2 days of enrollment
  The missed appointment proportion is based on the one appointment for which patients were contacted to receive a free ride

SECONDARY OUTCOMES:
Arrival time to clinic relative to the scheduled time (both arms) | Within 2 days of enrollment
Post-intervention, utilization frequency of acute care settings (both arms) | 7-days, 30-days, and 6 months post-appointment
Post-intervention, utilization frequency of primary care (both arms) | 7-days, 30-days, and 6 months post-appointment
Post-intervention, frequency of missed primary care appointments (both arms) | 30-days and 6-months post-appointment

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Internal Medicine Primary Care Practice, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chaiyachati KH, Hubbard RA, Yeager A, Mugo B, Lopez S, Asch E, Shi C, Shea JA, Rosin R, Grande D. Association of Rideshare-Based Transportation Services and Missed Primary Care Appointments: A Clinical Trial. JAMA Intern Med. 2018 Mar 1;178(3):383-389. doi: 10.1001/jamainternmed.2017.8336. PMID 29404572
- [Result] Chaiyachati KH, Hubbard RA, Yeager A, Mugo B, Shea JA, Rosin R, Grande D. Rideshare-Based Medical Transportation for Medicaid Patients and Primary Care Show Rates: A Difference-in-Difference Analysis of a Pilot Program. J Gen Intern Med. 2018 Jun;33(6):863-868. doi: 10.1007/s11606-018-4306-0. Epub 2018 Jan 29. PMID 29380214